CLINICAL TRIAL: NCT04937088
Title: Outpatient, Liquid Aspirin to Reduce COVID-19 Hospitalizations
Brief Title: Outpatient Liquid Aspirin (OLA)
Acronym: OLA COVID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Innovate Anti-Infectives (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: 1658
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Phase 2, proof of concept study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo and ASA 150 will be labeled to maintain blinding. The Principal Investigator and one Biostatistician will remain blinded to prevent any bias. Study staff/healthcare providers distributing the treatments to study subjects will be blinded to treatment assignment. Subjects will also be blinded to their treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Soy Bean Oil identical packaging as the active arm, taken once daily by mouth for 30 days.
  Interventions: Drug: ASA
- Liquid ASA (Active Comparator): Aspirin 150 mg liquid formulation (2.5%w/w) taken once daily by mouth for 30 days
  Interventions: Drug: ASA

INTERVENTIONS:
Drug: ASA — Liquid aspirin formulation

SUMMARY:
The purpose of this study is to obtain reliable and interpretable data to inform future trials regarding our hypothesis that a novel, liquid aspirin formulation can mitigate COVID -19 associated coagulopathy (CAC) . The potential impact is to reduce COVID-19 related hospitalization within 30 days of diagnosis due to (1) pulmonary events including respiratory failure; (2) cardiac events including myocardial infarction and myocarditis (3) venous or arterial thrombotic events; (4) acute renal insufficiency or failure.

DETAILED DESCRIPTION:
200 people will take part in this LSUHSC-NO and its affiliates study.

The clinical site will offer study enrollment to newly diagnosed COVID-19 patients at the time of diagnosis. Contact information will be shared with study team in a HIPAA compliant manner on the same day. Within 24 hours, our Study staff will contact patient for recruitment and enrollment. Within 48 hours of enrollment, the patient will come to a study site for randomization to treatment arms, to be provided a no-cost supply of the treatment which they are assigned, and for blood draws that help determine their risk of developing severe COVID disease. Patients will be assigned to either:

Arm 1: Placebo

Or

Arm 2: Treatment with liquid aspirin 150 mg daily. (ASA 150).

Study staff will follow-up every 2 days for a total of 30 days by text/phone/telemedicine to monitor changes in their health status, hospitalization rates, and encourage adherence to the treatment arm. Between days 7 and 10 of the study, patients will undergo repeat blood draws to help ensure their safety with regards to COVID-19. If they become hospitalized due to COVID-19, their participation will extend until they are discharged from the hospital. Medical records will be reviewed to collect data including demographics, medical comorbidities, laboratory data and hospitalization course. After 30 days of treatment, weekly follow up for another 30 days will take place ensure no late, adverse events occurred.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 40 years
* Written informed consent
* New (within 24 hours) COVID-19 diagnosis
* Serum 25OHD levels drawn at time of COVID-19 laboratory workup

Exclusion Criteria:

* Asymptomatic patients
* Patients already taking ASA and other anti-coagulant / anti-platelet therapies including but not limited to clopidogrel, heparin, low molecular weight heparin, coumadin, apixaban.
* Pregnant patients or prisoners
* History of GI bleeding or peptic ulcer disease, or spontaneous bleeding from other sites
* Thrombocytopenia (platelets <130,000/uL) at time of COVID diagnosis
* Anemia at time of COVID diagnosis (defined as hemoglobin level <12 g/dl in men or <11 g/dl in women)22
* History of chronic kidney disease
* Concurrent use of nonsteroidal anti-inflammatory drugs, or steroids
* Hypervitaminosis D and associated risk factors: Renal failure, Liver failure, Hyperparathyroidism, Sarcoidosis, Histoplasmosis
* Known allergy to Aspirin
* Inability to tolerate oral medications
* Known history of aspirin-induced asthma
* History of bleeding problems
* Patients who cannot avoid drinking 3 or more alcoholic drinks every day during the 30-day course of ASA treatment
* Patients who cannot stop taking other nonprescription NSAIDs (ibuprofen, naproxen, or others) during the 30-day course of ASA treatment
* Patients requiring hospitalization (for any reason) at time of screening
* Patients taking or who plan to take on an outpatient basis remdisivir, dexamethasone, or other therapies for treatment of COVID

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-12-05 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
Reduced COVID-19 related hospitalizations | 6 months
  To obtain reliable and interpretable data to inform future trials regarding our hypothesis that a 30 day treatment course of COVID patients with a novel, liquid aspirin formulation can reduce hospitalizations driven by COVID associate coagulopathy (CAC)

CONTACTS AND LOCATIONS:
Locations (1):
- Lsuhsc-No, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818